CLINICAL TRIAL: NCT05479526
Title: Investigation of the Effect of Tissue Properties of The Superficial Back Line on the Development of Plantar Fasciitis-Case Control Study
Brief Title: Effect of The Superficial Back Line on the Development of Plantar Fasciitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ayca Evkaya Acar, Lecturer, Istanbul Medeniyet University
Other Study IDs: 2022/0345
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Plantar Fascitis
Keywords: Plantar Fascitis; Fascia; Superficial Back Line

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Control group will consist of 42 healthy individuals, aged between 30-60 years.
- Group 2: This group will consist of 42 patients with diagnosed Plantar Fasciitis, aged between 30-60 years.

SUMMARY:
The primary aim of the study is to determine whether deviations from normal in the myofascial structure have an effect on the development of plantar fasciitis by evaluating the myofascial chain lines as well as the general evaluation parameters in patients diagnosed with plantar fasciitis. The secondary aim of the study is to create a future clinical projection regarding the applications to be made over the myofascial chain in addition to the generally accepted treatment protocols in the light of the findings.

DETAILED DESCRIPTION:
The plantar fascia is an important connective structure that extends from the metatarsal heads to the calcaneus and provides the continuity of the longitudinal arch of the foot. With microtraumas and the formation of chronic inflammation on the plantar surface exposed to repetitive stress, the fascia thickens and becomes prone to repetitive injuries and forms plantar fasciitis. The reasons for this repetitive stress are; excessive physical activity, obesity, age, prolonged standing, biomechanical changes, limited dorsiflexion and hamstring tension.

Studies on this subject in the literature have reported that tension in the hind leg muscles is associated with plantar fasciitis, and it has been shown that applications on the Achilles tendon and gastrocnemius relieve plantar fasciitis complaints. Similarly, it has been reported that tension in the hamstring muscle may be associated with the development of plantar fasciitis.

It is known that the Plantar Fascia and Achilles tendon affect each other due to the fascial connection, and therefore these structures are considered together in the solution of their problems. On the other hand, according to the fascial meridian concept developed by Thomas Myers, it was stated that the fascial connection between these two tissues extends to the frontal region in a chain manner, and that a problem at any point in the chain may cause problems in other elements of the chain. For this reason, recently, applications related to the detection and solution of problems have come to the fore by looking at fascial problems more holistically over the fascial chain.

Plantar Fascia; It is located in the Superficial Back Line and as far as we know, there is no plantar fasciitis study in which the myofascial chain is considered as a whole. Based on this, our aim in this study is to examine patients diagnosed with plantar fasciitis in terms of myofascial chain lines as well as general evaluation methods, to determine whether deviations from normal in the myofascial structure have an effect on the development of plantar fasciitis. Our main goal is to create projections for future clinical studies regarding the applications to be made over the myofascial chain in the treatment of plantar fasciitis in the light of the findings we have obtained.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers between the ages of 30-60
* Having experienced pain due to plantar fasciitis for at least 6 months
* Not having received medical treatment and/or physiotherapy for plantar fasciitis in the last 3 months.
* The participants' definition of pain over 3 according to the Visual Analogue Scale in the first step of the morning and this pain decreases with movements

Exclusion Criteria:

* Having history of lower extremity surgery and fracture in the last 6 months
* Having additional orthopedic, neurological and rheumatological diseases that may cause biomechanical malalignment, loss of muscle strength, and deterioration of gait parameters in the lower extremities, vertebral column and pelvis
* Having static foot deformity
* Having connective tissue disease that will affect tissue properties
* Having metabolic syndromes that may affect tissue properties such as diabetes
* Using sedatives and/or muscle relaxants that may alter muscle tone.
* Being diagnosed with obesity (BMI>30)
* Pregnancy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In the study, which is planned as a case-control study, the case group will consist of patients diagnosed with Plantar fasciitis, and the control group will consist of healthy people in the similar age group. The control group will consist of relatives of patients who meet the inclusion criteria and agree to participate in the study.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasonography | Baseline
  It will be used to measure the thickness of the plantar fascia. As a result of these studies, a plantar fascia greater than 4 mm appears to be abnormal and associated with plantar fasciitis. Ultrasonography (USG) evaluation is a routine method for the diagnosis of Plantar Fasciitis.
Plantar Fasciitis Pain | Baseline
  Visual Analogue Scale will be used in the assessment of pain severity. It expresses pain severity between a score of 0 (no pain) and 10 (unbearably severe pain)
Pes planus | Baseline
  Pes Planus will be evaluated with navicular drop test. The distance between the navicular bone and the ground is measured while the individual sits on the chair with the hip-knee joint in 90º flexion and the subtalar joint in neutral position. Then, the distance between the navicular bone and the ground is measured again while the individual is standing in a position with equal weight on both extremities. The difference between the two measurements is recorded. 10 mm or more difference is considered pes planus.
Foot Posture | Baseline
  Foot posture will be evaluated using the Foot posture index, a six item foot posture assessment tool, where each item is scored between -2 and +2 to give a sum total between -12 (highly supinated) and +12 (highly pronated). Items include: talar head palpation, curves above and below the lateral malleoli, calcaneal angle, talonavicular bulge, medial longitudinal arch, and forefoot to rearfoot alignment.
Ankle Joint Angle | Baseline
  Active and passive dorsi and plantar flexion angles will be measured with a goniometer.
Algometer | Baseline
  It is used to measure the pressure pain threshold. After localization of the painful area by palpation, force is applied with an algometer until patients feel pain and discomfort. The digit displayed on the algometer is recorded. The average of 3 measurements is taken.
Passive Tone | Baseline
  Passive Tone will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Stiffness | Baseline
  Stiffness will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Decrement | Baseline
  Decrement will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Creep | Baseline
  Creep will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Relaxation time | Baseline
  Relaxation time will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Hamstring Muscle shortness | Baseline
  Hamstring length will be measured with the straight leg lift test. The patient is asked to keep the opposite leg fixed on the bed with the knee straight in the supine position, wearing suitable clothes, and to raise the leg to be tested upwards with the ankle in dorsiflexion and the knee straight. The patient is instructed to wait where the initial tension occurs, and the last degree of movement is measured.
Pelvic tilt | Baseline
  The position of the pelvis will be evaluated with a digital pelvic inclinometer device to determine whether the pelvis has tilted anteriorly or posteriorly. The digital pelvic inclinometer is a valid and reliable method for the evaluation of pelvic tilt. The device consists of two calipers and the calipers are placed on the spina iliaca anterior superior (SIAS) and spina iliaca posterior superior (SIPS) of the pelvis. The score on the digital display is recorded. "-" values indicate posterior pelvic tilt, "+" values indicate anterior pelvic tilt.
Cervical and Lumbar Lordosis | Baseline
  It will be determined by photographing. Side photos will be taken while the patient is standing in a free standing position in front of a bare, flat wall with the upper body. Later, the obtained photo shoots will be analyzed with the Tracker 4.11.0 (Physlets, 2017) program and cervical and lumbar lordosis angles will be determined.
Skin temperature of the Plantar Fascitis area | Baseline
  In order to see the effectiveness of the applications, the skin temperature will be determined by thermal imaging method. This method is frequently preferred because it is a reliable and non-invasive method. The skin temperature of the plantar fascia will be measured with the P45 thermographic camera (Flir System, ThermaCAM, Sweden) with high thermal sensitivity, while the patient is in the prone position, while the feet are hanging from the bed at the level of the malleolus. The measurement will be made by placing the camera on a tripod placed 1m away from the patient. In the analysis, the area covering 1 cm distance from the point where fasciitis develops will be used. Skin temperature will be determined using the FLIR Quick-Report 1.2 software, one of the temperature indicators obtained from this region. In the calculation of skin temperature, the human skin emissivity value will be accepted as 0.98.
Headache | Baseline
  Presence of headache will be questioned and severity assessment will be made with Visual Analogue Scale. It expresses pain severity between a score of 0 (no pain) and 10 (unbearably severe pain).
Windlass Test | Baseline
  While the patient is sitting in a chair, the big toe of the foot to be tested is brought into the dorsal flexion of the metatarsal phalangeal joint for a hard time. Pain at the junction of the plantar fascia with the calcaneus during this movement indicates a positive test.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Kablan, Asst. Prof., Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arshad Z, Aslam A, Razzaq MA, Bhatia M. Gastrocnemius Release in the Management of Chronic Plantar Fasciitis: A Systematic Review. Foot Ankle Int. 2022 Apr;43(4):568-575. doi: 10.1177/10711007211052290. Epub 2021 Nov 12. PMID 34766860
- [Background] Hoefnagels EM, Weerheijm L, Witteveen AG, Louwerens JK, Keijsers N. The effect of lengthening the gastrocnemius muscle in chronic therapy resistant plantar fasciitis. Foot Ankle Surg. 2021 Jul;27(5):543-549. doi: 10.1016/j.fas.2020.07.003. Epub 2020 Jul 12. PMID 32773360
- [Background] Lee JH, Jung HW, Jang WY. A prospective study of the muscle strength and reaction time of the quadriceps, hamstring, and gastrocnemius muscles in patients with plantar fasciitis. BMC Musculoskelet Disord. 2020 Nov 5;21(1):722. doi: 10.1186/s12891-020-03740-1. PMID 33153452